CLINICAL TRIAL: NCT02585895
Title: A Randomized, Actively Controlled, Open-label, Multicenter Study of Efficacy and Safety of Evolocumab Compared With Low Density Lipoprotein Cholesterol (LDL-C) Apheresis, Followed by Single-Arm Evolocumab Administration in Subjects Receiving LDL-C Apheresis Prior to Study Enrollment
Brief Title: Evolocumab Compared to LDL-C Apheresis in Patients Receiving LDL-C Apheresis Prior to Study Enrollment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140316; 2015-001343-37 (EudraCT Number)
Record Dates: First submitted 2015-10-07; First posted 2015-10-26 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Hypercholesterolemia
Keywords: LDL-C Apheresis; Hypercholesterolemia; Elevated Cholesterol; High Cholesterol; PCSK9 mutations; Severe Familial Hypercholesterolemia; evolocumab; Repatha
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipoproteinemia Type II | interventions — evolocumab; Cholesterol, LDL; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Evolocumab (Experimental): Participants received 140 mg evolocumab every 2 weeks (Q2W) administered by subcutaneous injection for 6 weeks during the primary period of the study. Starting at week 6 (beginning of the post-primary period), participants received 140 mg evolocumab Q2W up to week 24.
  Interventions: Biological: Evolocumab
- Low Density Lipoprotein Cholesterol (LDL-C) Apheresis (Active Comparator): Participants continued apheresis at the same schedule, every week (QW) or every two weeks (Q2W), as prior to study entry, for the first 6 weeks. Starting at week 6 (beginning of the post-primary period), participants received 140 mg evolocumab Q2W up to week 24.
  Interventions: Biological: Evolocumab; Procedure: Low-density Lipoprotein Cholesterol (LDL-C) Apheresis

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection once every 2 weeks
  Other Names: Repatha; AMG 145
Procedure: Low-density Lipoprotein Cholesterol (LDL-C) Apheresis — Participants received apheresis for LDL-C according the their physician's prescription and local custom.
  Arms: Low Density Lipoprotein Cholesterol (LDL-C) Apheresis

SUMMARY:
To evaluate the efficacy of subcutaneous (SC) evolocumab, compared to regularly scheduled low-density lipoprotein cholesterol (LDL-C) apheresis, on reducing the need for future apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age
* Subject has been receiving regular apheresis for LDL-C lowering for at least 3 months immediately prior to lipid screening and has a treatment goal of LDL-C < 100 mg/dL (2.6 mmol/L), and has been receiving LDL-C apheresis during the last ≥ 4 weeks prior to lipid screening at regular QW or Q2W schedule and with no changes in apheresis type
* Subject is receiving lipid-lowering pharmacological background therapy which includes a high-intensity statin dose (moderate-intensity statin dose with attestation that a higher dose is not appropriate for the subject) unless the subject has a history of statin intolerance
* Lipid-lowering therapy status (ie, any therapy for lowering lipids, including apheresis type and frequency) must be unchanged for ≥ 4 weeks prior to LDL-C screening
* Pre-apheresis LDL-C is ≥ 100 mg/dL (≥ 2.6 mmol/L) and ≤ 190 mg/dL (≤ 4.9 mmol/L) at screening
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L) at screening.

Exclusion criteria:

* Known homozygous familial hypercholesterolemia
* Missing any apheresis session is medically contraindicated or inappropriate
* Stopping apheresis would be inappropriate in the opinion of the investigator even if LDL-C is controlled to < 100 mg/dL with other therapies
* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months prior to randomization.
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-12-21 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (4):
  - Research Site, Boca Raton, Florida
  - Research Site, Kansas City, Kansas
  - Research Site, Grandville, Michigan
  - Research Site, Portland, Oregon
- Research Site, Heidelberg, Victoria, Australia
- Research Site, Hradec Králové, Czechia
- France (2):
  - Research Site, Bron
  - Research Site, Nantes
- Germany (4):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Flensburg
- Italy (2):
  - Research Site, Pisa
  - Research Site, Roma
- Research Site, Seville, Andalusia, Spain
- United Kingdom (2):
  - Research Site, Harefield
  - Research Site, Penarth

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Baum SJ, Sampietro T, Datta D, Moriarty PM, Knusel B, Schneider J, Somaratne R, Kurtz C, Hohenstein B. Effect of evolocumab on lipoprotein apheresis requirement and lipid levels: Results of the randomized, controlled, open-label DE LAVAL study. J Clin Lipidol. 2019 Nov-Dec;13(6):901-909.e3. doi: 10.1016/j.jacl.2019.10.003. Epub 2019 Oct 11. PMID 31759938
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 15 centers in the following 8 countries: Australia, Czech Republic, France, Germany, Italy, Spain, the United Kingdom, and the United States. Participants were enrolled from 21 December 2015 to 21 July 2016.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to continue apheresis on the same schedule as before study entry, or to stop apheresis and receive evolocumab. Randomization was stratified by screening low-density lipoprotein cholesterol (LDL-C) (< 160 mg/dL [4.1 mmol/L] vs ≥ 160 mg/dL).
Groups:
- Apheresis: Participants continued apheresis at the same schedule, every week (QW) or every two weeks (Q2W), as prior to study entry, for the first 6 weeks. Starting at week 6 (beginning of the post-primary period), participants received 140 mg evolocumab Q2W up to week 24.
Period: Primary Period
Arm/Group | Apheresis | Evolocumab
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0
Period: Post-primary Period
Arm/Group | Apheresis | Evolocumab
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apheresis | Evolocumab | Total
Number analyzed (Participants) | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.0) | 65.4 (8.1) | 62.4 (9.5)
Age, Customized [Number; unit: participants]
  < 65 years | 14 | 7 | 21
  ≥ 65 years | 6 | 12 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 13 | 10 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 20 | 18 | 38
Stratification Factor: Screening LDL-C Level [Number; unit: participants]
  < 160 mg/dL | 11 | 11 | 22
  ≥ 160 mg/dL | 9 | 8 | 17
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] | 150.6 (25.6) | 152.4 (21.2) | 151.5 (23.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Apheresis Avoidance at the End of Randomized Therapy
Description: Avoidance of apheresis at end of randomized therapy was defined as no apheresis at week 5 and week 6. Aperesis at weeks 5 or 6 was based on LDL-C level at week 4:
  participants with LDL-C ≥ 100 mg/dL at week 4 received apheresis at week 5 (participants who received apheresis QW before study entry) or week 6 (participants who received apheresis Q2W prior to study entry). If LDL-C was < 100 mg/dL at week 4, no apheresis was performed at week 5 or week 6, irrespective of assigned treatment group.
  Participants who ended the study prior to week 6 were considered as not achieving apheresis avoidance.
Time Frame: Week 5 and week 6
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apheresis | Evolocumab
Number analyzed (Participants) | 20 | 19
percentage of participants | 10.0 [2.8 to 30.1] | 84.2 [62.4 to 94.5]
Statistical Analysis 1: Comparison: Apheresis vs Evolocumab; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Based on Cochran-Mantel-Haenszel (CMH) test stratified by screening LDL-C level; Treatment Difference = 74.2, 95% CI 2-sided [44.6 to 86.8] — Treatment difference used apheresis as the reference

2. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol
Time Frame: Baseline and week 4
Population: Randomized participants with non-missing data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Apheresis | Evolocumab
Number analyzed (Participants) | 19 | 19
percent change | 2.61 (3.97) | -50.13 (4.03)
Statistical Analysis 1: Comparison: Apheresis vs Evolocumab; Test type: Superiority or Other; p < 0.0001, Repeated measures linear effects model; Model included treatment group, screening LDL-C level, scheduled visit, and the interaction of treatment group with scheduled visit as covariates; Treatment Difference = -52.74, 95% CI 2-sided [-64.18 to -41.30], Standard Error of Mean 5.64 — Treatment difference used apheresis as the reference

3. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein-Cholesterol
Time Frame: Baseline and Week 4
Population: Randomized participants with non-missing data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Apheresis | Evolocumab
Number analyzed (Participants) | 19 | 19
percent change | 1.80 (3.29) | -44.58 (3.34)
Statistical Analysis 1: Comparison: Apheresis vs Evolocumab; Test type: Superiority or Other; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; Treatment Difference = -46.37, 95% CI 2-sided [-55.85 to -36.90], Standard Error of Mean 4.67 — Treatment difference used apheresis as the reference

4. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/High-density Lipoprotein Cholesterol Ratio
Time Frame: Baseline and Week 4
Population: Randomized participants with non-missing data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Apheresis | Evolocumab
Number analyzed (Participants) | 19 | 19
percent change | 0.15 (2.65) | -35.65 (2.67)
Statistical Analysis 1: Comparison: Apheresis vs Evolocumab; Test type: Superiority or Other; p < 0.0001, Repeated measures linear effects model; [statistical method as in outcome 2, analysis 1]; Treatment Difference = -35.80, 95% CI 2-sided [-43.39 to -28.21], Standard Error of Mean 3.74

ADVERSE EVENTS:
Time Frame: 6 weeks during the primary period and 20 weeks during the post-primary period.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Primary Period: Apheresis QW: Participants received apheresis every week (QW) for 6 weeks during the primary period of the study.
- Primary Period: Apheresis Q2W: Participants received apheresis every 2 weeks (Q2W) for 6 weeks during the primary period of the study.
- Primary Period: Evolocumab: Participants received 140 mg evolocumab every 2 weeks (Q2W) administered by subcutaneous injection for 6 weeks during the primary period of the study.
- Post-primary Period: Apheresis/Evolocumab: Starting at week 6 participants received 140 mg evolocumab Q2W up to week 24.
- Post-primary Period: Evolocumab/Evolocumab: Participants received 140 mg evolocumab Q2W from week 6 to week 24.
Arm/Group | Primary Period: Apheresis QW | Primary Period: Apheresis Q2W | Primary Period: Evolocumab | Post-primary Period: Apheresis/Evolocumab | Post-primary Period: Evolocumab/Evolocumab
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/16 | 0/19 | 0/20 | 2/19
Other Adverse Events (participants affected / at risk) | 2/4 | 5/16 | 10/19 | 6/20 | 8/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Period: Apheresis QW (N=4) | Primary Period: Apheresis Q2W (N=16) | Primary Period: Evolocumab (N=19) | Post-primary Period: Apheresis/Evolocumab (N=20) | Post-primary Period: Evolocumab/Evolocumab (N=19)
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Period: Apheresis QW (N=4) | Primary Period: Apheresis Q2W (N=16) | Primary Period: Evolocumab (N=19) | Post-primary Period: Apheresis/Evolocumab (N=20) | Post-primary Period: Evolocumab/Evolocumab (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 2 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Mastitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 2 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Menopause (Social circumstances) | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.